CLINICAL TRIAL: NCT01724554
Title: A Single-center, Open-label Study Evaluating the Impact of Repeat Intravitreal Injections of Aflibercept on Capillary Non-Perfusion (CNP) in Subjects With Proliferative Retinopathy and/or Macular Edema Secondary to Proliferative Diabetic Retinopathy and Central Retinal Venous Occlusive Disease
Brief Title: Impact of Intravitreal Aflibercept Injections on Capillary Non-Perfusion
Acronym: ANDROID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ophthalmic Consultants of Boston (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANDROID
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Central Retinal Vein Occlusion; Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Every Month Treatment (Experimental): Patients will receive Intravitreal Aflibercept Injection (IAI) every month for the 12 month duration of the study.
  Interventions: Drug: Intravitreal Aflibercept Injection
- Every Month, then Every Other Month (Experimental): Patients will receive Intravitreal Aflibercept Injection (IAI) every month for the first 6 months, then every other month for the next 6 months. Retreatment criteria will allow for patients to be treated every month in the second 6 months if needed.
  Interventions: Drug: Intravitreal Aflibercept Injection

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection — Aflibercept administered to the eye intravitreally either every month or every other month.
  Other Names: IAI

SUMMARY:
The purpose of this study is to look at how effective, safe, and well tolerated Intravitreal Aflibercept Injection is in subjects with Central Retinal Vein Occlusion (CRVO) or Proliferative Diabetic Retinopathy (PDR).

DETAILED DESCRIPTION:
Protocol available upon request.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of one or more of the following:

   Proliferative retinopathy (PDR) Macular edema secondary to CRVO Proliferative disease secondary to CRVO (anterior segment or posterior segment neovascularization).
2. Be in need of IAI treatment, whether previously treated or treatment-naïve.
3. Age > 18 years.

Exclusion Criteria:

1. Subjects with macular edema secondary to diabetic retinopathy without concomitant proliferative diabetic retinopathy.
2. Subjects with cataract or other media opacities impairing adequate visualization of the retina to the extent that good quality images are impossible.
3. Presence of any substantial ocular disease (other than diabetic retinopathy or central retinal vein occlusion) that may compromise vision in the study eye and /or confound interpretation of the data; e.g. substantial cataracts, advanced glaucoma, optic neuritis, optic neuropathy or atrophy, marked macular atrophy, history of retinal detachment, uveitis, viral or other forms of chorioretinitis, etc.
4. Active intraocular inflammation (grade trace or above) in the study eye, or history of idiopathic or autoimmune-associated uveitis in either eye.
5. Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication).
6. History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye.
7. Participation in a study of an investigational drug or device within 30 days prior to potential enrollment into the study.
8. Intraocular surgery (including cataract surgery) in the study eye within 60 days preceding baseline.
9. History of vitrectomy surgery in the study eye.
10. Subjects with 12 or more anti-VEGF injections within 24 months prior to Screening.
11. Subjects who received anti-VEGF therapy within 30 days of Screening or received steroid or laser therapy within 90 days of Screening.
12. Subjects allergic to fluorescein, povidone iodine (Betadyne) or aflibercept
13. Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Mean Change in Capillary Non-Perfusion | 12 months
  To determine mean change in the presence and amount of capillary non-perfusion as measured by wide-angle angiography using Optos 200Tx system at Baseline, Month 3, Month 6, and Month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States